CLINICAL TRIAL: NCT07347249
Title: A Clinical Study to Assess the Safety and Efficacy of Sutacimig in Participants With Congenital Factor VII Deficiency
Brief Title: A Clinical Study to Assess Sutacimig in Participants With Congenital Factor VII Deficiency
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hemab ApS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMB-001-201
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Congenital Factor VII Deficiency
Keywords: Congenital Factor VII Deficiency; Factor VII Deficiency; FVIID; Congenital coagulation factor VII (FVII) deficiency
MeSH Terms: conditions — Factor VII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with a FVII(a) level of < 10% (Experimental)
  Interventions: Drug: Sutacimig
- Participants with a FVII(a) level of ≥10% (Experimental)
  Interventions: Drug: Sutacimig

INTERVENTIONS:
Drug: Sutacimig — Sutacimig is a subcutaneously administered, bispecific antibody being developed as a prophylactic treatment option for congenital bleeding disorders.
  Arms: Participants with a FVII(a) level of < 10%
Drug: Sutacimig — Sutacimig is a subcutaneously administered, bispecific antibody being developed as a prophylactic treatment option for congenital bleeding disorders.
  Arms: Participants with a FVII(a) level of ≥10%

SUMMARY:
Open-label study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of a single dose of sutacimig monotherapy in participants with congenital FVII deficiency (FVIID).

DETAILED DESCRIPTION:
The objective is to administer a single dose of sutacimig and to evaluate safety, pharmacokinetics, and pharmacodynamics. Two cohorts may be evaluated. Cohort A is defined by participants with a FVII(a) level of < 10%. Cohort B is defined by participants with a FVII(a) level of ≥10%.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years, inclusive, at the time of signing informed consent.
2. Diagnosis of FVIID defined by Factor VII:C activity < 10% documented on ≥ 2 different laboratory measurements by local laboratory assessment.
3. Severe bleeding history characterized by history of a major bleeding event and/or receipt of recombinant activated FVII or fresh frozen plasma as treatment for bleeding or a severe clinical bleeding history as defined by the Investigator.
4. Has the ability to provide informed consent to participate in the trial.

Exclusion Criteria:

1. Presence of known inhibitors to FVII or FVIIa
2. History of clinically significant hypersensitivity associated with monoclonal antibody therapies.
3. History of venous or arterial thrombosis or thromboembolic disease, with the exception of catheter-associated superficial vein thrombosis.
4. Known thrombophilia risk by the following criteria: Homozygous Factor V Leiden (FVL), compound heterozygous FVL/Prothrombin gene mutation, antithrombin <50%, congenital protein C, and protein S deficiency with levels <50%.
5. Clinically significant comorbidity that may interfere with study participation.
6. Use of concomitant therapy not permitted during the study (i.e., other platelet inhibitors, desmopressin, fibrinolysis inhibitors, except if used as local treatment [e.g., for oral bleeds])
7. Female participants who are pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 through Day 57

SECONDARY OUTCOMES:
Pharmacokinetic Parameter: Maximum observed plasma concentration (Cmax) of sutacimig | Day 1 through Day 57
Pharmacokinetic Parameter: Time to reach maximum observed plasma concentration (Tmax) | Baseline through Day 57
Pharmacokinetic Parameter: Area under the plasma concentration-time curve from time zero to last quantifiable concentration (AUClast) | Day 1 through Day 57
Pharmacokinetic Parameter: Area under the curve from time zero to extrapolated infinite time (AUCinf) | Day 1 through Day 57
Pharmacokinetic Parameter: Terminal elimination phase half-life (T1/2) | Day 1 through Day 57
Pharmacodynamic Parameter: Total Factor VII | Day 1 through Day 57
Pharmacodynamic Parameter: Factor VII Activity | Day 1 through Day 57
Pharmacodynamic Parameter: Prothrombin time (PT) Measurement | Day 1 through Day 57
Pharmacodynamic Parameter: Activated partial thromboplastin time (aPTT) Measurement | Day 1 through Day 57
Anti-drug antibody levels | Day 1 through Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor Website — https://www.hemab.com/